CLINICAL TRIAL: NCT04584801
Title: A Comparative, Multi Centre Study, to Develop a Model for Structured Light Plethysmography Against Standard of Care in the Diagnosis of Chronic Obstructive Pulmonary Disease for Patients Who Plan to Undergo Spirometry Testing
Brief Title: SLP Model Development in the Diagnosis of COPD Patients
Acronym: SLPCOPD
Status: Completed | Type: Observational
Sponsor: Pneumacare Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: PMC-SLPCOPD-2020
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-01

CONDITIONS: COPD; Healthy Smoker
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- COPD Patients: Development Phase Any adult (≥18 years old) who has been diagnosed with COPD guide GOLD criteria (FEV1/FVC ratio post bronchodilator <0.70)
  * Cohort A (N=50): COPD stage 1
  * Cohort B (N=50): COPD stage 2
  * Cohort C (N=50): COPD stage 3
  * Cohort D (N=50): COPD stage 4
  Interventions: Device: Structured Light Plethysmography
- Healthy Smoker Subjects: • Cohort E (N=50): Healthy Smokers (≥35 years old, current or ex-smoker with a history of ≥10 pack-years (20 cigarettes smoked per day for 1 year)
  Interventions: Device: Structured Light Plethysmography

INTERVENTIONS:
Device: Structured Light Plethysmography — Development Phase (Original Part A): Participants will have two 5-minute SLP measurements (Pre and Post bronchodilator).
  Participants will also undergo standard of care spirometry assessment
  Other Names: Thora-3Di™

SUMMARY:
This is an observational, comparative, multicentre study to develop a model for the Thora3Di™ against standard practice in patients who are undergoing investigation for COPD. The core methodology involves capturing of data during a short period of measurement of breathing using SLP against spirometric outcomes.

DETAILED DESCRIPTION:
This study will generate data to characterise the tidal breathing patterns and parameters with Thora-3Di™ against spirometry FEV1/FVC and %predicted. Subjects will have a Part A visit (Development Phase) to develop algorithms for COPD diagnosis. At Part A visit, subjects will have two 5-minute SLP measurements (Pre and Post bronchodilator). The SLP measurement should be performed prior to standard lung function tests with minimal impact on clinical time and no change to hospital attendance. Also, subjects will be asked to report concomitant medications and adverse events and fill in COPD assessment test (CAT™).

ELIGIBILITY:
Inclusion Criteria:

* Any adult (≥18 years old) who has been diagnosed with COPD guide GOLD criteria (FEV1/FVC ratio post bronchodilator <0.70)
* Healthy Smokers (≥35 years old, current or ex-smoker with a history of ≥10 pack years (20 cigarettes smoked per day for 10 year))

Exclusion Criteria:

* Be unable to sit in an upright position for required period
* Have had deteriorated COPD symptoms since the last spirometry unless willing to undergo spirometry testing
* Have significant co-morbidities (i.e. Chest work or spinal deformity, OSA, AHI >30 secs
* Any other significant disease or disorder which, in the opinion of the investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participants' ability to participate in the study
* Height > 194 cm
* BMI >40
* Female participant who is pregnant, lactating or planning pregnancy during the course of the study
* Be unable to consent or comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Development Phase (Original Part A)
  * Cohort A (N=50): COPD stage 1
  * Cohort B (N=50): COPD stage 2
  * Cohort C (N=50): COPD stage 3
  * Cohort D (N=50): COPD stage 4
  * Cohort E (N=50): Healthy Smokers (≥35 years old, current or ex-smoker with a history of ≥10 pack-years (20 cigarettes smoked per day for 1 year)
Sampling Method: Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
To develop a machine learning model to use SLP data in patients diagnosed with COPD or healthy smokers to predict historical spirometry results (within 6 months) or prospective spirometry results, and classify subjects according to COPD/non-COPD. | 2 years
  The proportion of points falling between the upper and lower 95% CIs of the Bland-Altman plot of the average of FEV1/FVC spirometer values and the output from the model using the SLP parameters against the difference between the spirometer values and their SLP parameter model counterparts.

SECONDARY OUTCOMES:
To evaluate the safety of the Thora-3Di™ | 2 years
  Incidence of adverse events while the SLP techniques are carried out.

CONTACTS AND LOCATIONS:
Overall Officials: Mona Bafadhel, PhD, Study Chair — King's College London; Dennis Wat, MD, Principal Investigator — Liverpool Heart and Chest Hospital NHS Trust; Brendan Cooper, PhD, Principal Investigator — University Hospital Birmingham NHS Foundation Trust; Paul Walker, MD, Principal Investigator — Liverpool University Hospital NHS Foundation Trust; Richa Singh, MD, Principal Investigator — London Barts Health NHS Foundation Trust; Mitra Shahidi, MD, Principal Investigator — Buckinghamshire Healthcare NHS Trust; Sanjay Ramakrishnan, MD, Principal Investigator — Oxford University Hospitals NHS Trust; Suraj Rajput, MSc, Principal Investigator — Medway Community Healthcare
Locations (7):
- United Kingdom (7):
  - Buckinghamshire Healthcare NHS Trust - Stoke Mandeville Hospital, Aylesbury
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Medway Community Healthcare, Gillingham
  - Liverpool Heart and Chest Hospital, Liverpool
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - Barts Health NHS Trust - the Royal London Hospital, London
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No
Via UK NIHR website